CLINICAL TRIAL: NCT04278066
Title: Hyper-Cardia Study : Hyperoxia and Pulmonary Complications After Cardiac Surgery
Brief Title: Hyperoxia and Pulmonary Complications After Cardiac Surgery
Acronym: HYPER-CARDIO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7655
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-02

CONDITIONS: Hyperoxia
Keywords: Hyperoxia; Cardiac surgery; pulmonary complications; Lung collapse; Post-operative
MeSH Terms: conditions — Hyperoxia; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to demonstrate that hyperoxia in cardiac surgery increase the occurrence of post-operative pulmonary complications

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Patient operated heart surgery with extra-corporal life support
* Hospitalization in Cardiology intensive and critical care unit
* Patient operated in HUS between 01/01/2015 and 31/12/2019
* Subject consent, after information, to the reuse of its data for the purposes of this study

Exclusion Criteria:

* Non-consent patient
* Hypoxemic patient
* Emergency surgery
* Patient with post-operative cardiac assist device
* Patient with guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient operated heart surgery with extra-corporal life support
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Retrospective study of the average of per and postoperative PaO2 in cardiac surgery | iles analyzed retrospectily from January 1st, 2015 to December 31, 2019 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: François FISCHER, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service d'Anesthésiologie - NHC, Strasbourg, France